CLINICAL TRIAL: NCT01768338
Title: A Phase I Study of Recombinant Human Interleukin-18 (SB-485232) in Combination With Ofatumumab After Autologous Peripheral Blood Stem Cell Transplantation for Lymphoma
Brief Title: Recombinant Human IL-18 and Ofatumumab After PBSCT for Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael John Robertson (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Michael John Robertson, Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUCRO-0397; 1210009882 (Other: Indiana University Institutional Review Board)
Record Dates: First submitted 2013-01-09; First posted 2013-01-15 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Interleukin-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ofatumumab combined with SB-485232 (Experimental): Otatumumab: 1000 mg IV for 4 weeks. SB-485232: escalating doses (3 ug/kg up to 30 ug/kg) for 8 weeks.
  Interventions: Drug: Ofatumumab combined with SB-485232

INTERVENTIONS:
Drug: Ofatumumab combined with SB-485232 — Ofatumumab with escalating doses of SB-485232

SUMMARY:
The purpose of this study is to test the safety of rhIL-18 combined with ofatumumab to see what effects (good and bad) it has on subjects and their non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone high-dose therapy and autologous PBSCT for treatment of CD20+ lymphoma.
* Patients must be between 2-6 months post-transplantation at the time of study registration.
* Patients must have at least stable disease (no overt progressive disease) at the time of study registration.
* Laboratory values must be within protocol specified ranges.
* Females of childbearing potential must have a negative pregnancy test.
* Females of childbearing potential and males must use an effective method of contraception from the time of consent until at least 365 days following discontinuation of protocol therapy.

Exclusion Criteria:

* Patient must not have obvious clinical progression of lymphoma after PBSCT as determined by the treating physician.
* Cannot be positive for hepatitis B surface antigen, hepatitis B core antibody or HIV antibody.
* No major or uncontrolled comorbid conditions as determined by the treating physician: history of ventricular arrhythmias requiring drug or device therapy; uncontrolled angina or symptomatic congestive heart failure; • severe or uncontrolled infection requiring systemic antibiotic or antifungal therapy or active hepatitis C infection; severe or uncontrolled psychiatric illness.
* No known leptomeningeal involvement by lymphoma or current metastatic brain disease.
* No Corrected QTc interval > 480 msec.
* No known or suspected hypersensitivity to ofatumumab or SB-485232 that in the opinion of the investigator is a contraindication to their participation in the study.
* No systemic (oral or parenteral) corticosteroids within 14 days of study entry.
* Not receiving concurrent chemotherapy, biologic therapy, radiotherapy, or other investigational therapy.
* No previous treatment with SB-485232 or ofatumumab.
* No history of other malignancy except for adequately treated non-invasive cancers of the skin (basal or squamous cell) or carcinoma in situ of the uterine cervix.
* No diabetes mellitus with poor glycemic control (documented hemoglobin A1c >7% within 4 weeks prior to study entry).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-02; Primary Completion 2016-03 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the the number of subjects with adverse events who receive SB-485232 when given in combination with ofatumumab | 8 weeks
  Adverse events will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0 which uses a scale of 1 (mild) to 5 (caused death).

SECONDARY OUTCOMES:
To evaluate the biologic effects of SB-485232 given in combination with ofatumumab | 8 weeks
  Biologic effects will be assessed by flow cytometric analysis of PBMCs and ELISA tests to measure plasma cytokines and chemokines.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Robertson, MD, Principal Investigator — Indiana University Melvin and Bren Simon Cancer Center
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No